CLINICAL TRIAL: NCT03477903
Title: A Phase 2b, Randomized, Multi-Center, Double-Blind, Dose-Ranging Study to Assess the Efficacy, Safety and Pharmacokinetics of Intravenous TAK-954 in Critically Ill Patients With Enteral Feeding Intolerance
Brief Title: TAK-954 in Critically Ill Participants With Enteral Feeding Intolerance (EFI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment; No safety concerns
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-954-2002; U1111-1208-1831 (Other: WHO); 2017-003206-41 (EudraCT Number); 18/NE/0139 (Registry Identifier: NRES)
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness; Enteral Nutrition; Enteral Feeding Intolerance
Keywords: Drug therapy
MeSH Terms: conditions — Critical Illness | interventions — Metoclopramide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: TAK-954 0.1 mg (Experimental): TAK-954 0.1 milligram (mg), intravenously, administered as 60 minute-infusion, once daily along with 2 milliliter (mL) normal saline injection, intravenously, three times a day for a minimum of 5 days up to a maximum of 14 days.
  Interventions: Drug: TAK-954; Drug: Normal Saline
- Group B: TAK-954 0.3 mg (Experimental): TAK-954 0.3 mg, intravenously, administered as 60 minute-infusion, once daily along with 2 mL normal saline injection, intravenously, three times a day for a minimum of 5 days up to a maximum of 14 days.
  Interventions: Drug: TAK-954; Drug: Normal Saline
- Group C: TAK-954 1.0 mg (Experimental): TAK-954 1.0 mg, intravenously, administered as 60 minute-infusion, once daily along with 2 mL normal saline injection, intravenously, three times a day for a minimum of 5 days up to a maximum of 14 days.
  Interventions: Drug: TAK-954; Drug: Normal Saline
- Group D: Metoclopramide 10 mg (Active Comparator): Metoclopramide 10 mg, injection, intravenously, three times a day along with 100 mL normal saline 60-minute infusion, intravenously, once daily for a minimum of 5 days up to a maximum of 14 days.
  Interventions: Drug: Metoclopramide; Drug: Normal Saline

INTERVENTIONS:
Drug: TAK-954 — TAK-954 infusion
  Arms: Group A: TAK-954 0.1 mg; Group B: TAK-954 0.3 mg; Group C: TAK-954 1.0 mg
Drug: Metoclopramide — Metoclopramide infusion
  Arms: Group D: Metoclopramide 10 mg
Drug: Normal Saline — 0.9% sodium chloride for injection

SUMMARY:
The purpose of this study is to assess the treatment effect of intravenous TAK-954 in improving the average daily protein adequacy received through enteral nutrition in critically-ill participants developing EFI.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. The study will assess the treatment effect of intravenous TAK-954 in improving average daily protein adequacy received through enteral nutrition in critically ill participants with EFI.

The study will enroll approximately 200 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the 4 treatment groups -which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Group A: TAK-954 0.1 mg
* Group B: TAK-954 0.3 mg
* Group C: TAK-954 1 mg
* Group D: Metoclopramide 10 mg

This multi-center trial will be conducted in the United States, United Kingdom, Australia and Canada. The overall duration of treatment in this study is maximum of 14 days while in hospital. Participants will be contacted by telephone 30 and 90 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has at least a size 12-(french size) Fr nasogastric or orogastric tube with its tip at least 10 centimeter (cm) below the esophagogastric junction confirmed radiologically (the tip of the tube must be in the body or the antrum of the stomach and not in the fundus).
2. Is intubated and mechanically ventilated in the ICU.
3. Is expected to remain alive, mechanically ventilated, and receive continuous enteral feeding for >=48 hours following randomization.
4. Have EFI, defined as a single GRV measurement of >=250 mL with vomiting/retching within the last 24 hours, or a single GRV measurement of >=500 mL with or without vomiting/retching within the last 24 hours.

Exclusion Criteria:

1. Is under consideration for withdrawal of life-sustaining treatments within the next 72 hours.
2. Has had major esophageal or gastric surgery or direct luminal trauma on this admission (participants with lower abdominal surgery are not excluded unless enteral feeding is contraindicated).
3. Has mechanical bowel obstruction, short bowel syndrome, or the presence of an active gastric pacemaker.
4. Have pre-existing hepatic disease that meets Child-Pugh Class B (moderate; total score 7 to 9 points) or C (severe; total score 10 to 15 points).
5. Has been admitted primarily for treatment of a drug overdose.
6. Has a presence of a post-pyloric tube in place at Randomization that may be used for enteral nutrition.
7. Is receiving parenteral nutrition (PN) at Screening.
8. Is in diabetic ketoacidosis or non-ketotic hyperosmolar coma.
9. Has a different nutrient requirement than allowed in feeding protocol.(outside a range of 1.2 to 2 gram per kilogram per day [g/kg/day] of proteins and up to 1.5 kilocalorie per milliliter [kcal/mL]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (44):
- United States (14):
  - Joseph M Still Burn Centers, Augusta, Georgia
  - Eastern Idaho Medical Consultants, Idaho Falls, Idaho
  - Illinois Lung & Critical Care Institute, Peoria, Illinois
  - University of Kentucky Health Care, Lexington, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Truman Medical Center Hospital Hill, Kansas City, Missouri
  - Creighton University, Omaha, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - New York-Presbyterian Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Froedtert Hospital, Wauwatosa, Wisconsin
- Australia (10):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Logan Hospital, Meadowbrook, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Northern Hospital, Epping, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Canada (7):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - Hopital Charles-LeMoyne, Greenfield Park, Quebec
  - Hopital du Sacre-Coeur de Montreal, Monteal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec Hospital Centre Hospitalier de IUniversite Laval, Québec, Quebec
- United Kingdom (13):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Royal Sussex County Hospital, Brighton, England
  - University Hospitals Bristol NHS Foundation Trust, Bristol, England
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - The Royal London Hospital, London, England
  - Royal Free London NHS Foundation Trust, London, England
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - NHS Lothian, Edinburgh, Scotland
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - Cardiff and Vale University Health Board, Cardiff, Wales
  - Aneurin Bevan University Health Board, Newport, Wales
  - Royal Liverpool University Hospital NHS Trust, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant took part in the study at an investigative site in the United States from 25-Aug-2018 to 29-Aug-2018.
Pre-assignment Details: One participant with a diagnosis of Enteral Feeding Intolerance (EFI) was enrolled and received 0.1 mg of TAK-954. No participants were enrolled in the other 3 planned arms of the study.
Groups:
- TAK-954 0.1 mg: TAK-954 0.1 milligrams (mg), intravenously, administered as 60 minute-infusion, once daily along with 2 milliliters (mL) normal saline injection, intravenously, three times a day for a minimum of 5 days up to a maximum of 14 days.
Period: Overall Study
Arm/Group | TAK-954 0.1 mg
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Region of Enrollment [Count of Participants; unit: Participants] — Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
  Participants
    United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Protein Adequacy Over the First 5 Days of Treatment
Description: Average daily protein adequacy received through enteral nutrition is defined as the percentage of goal protein delivered per day, where percentage of goal protein delivered is calculated as the ratio of actual protein achievement to the total participant-specific target protein prescribed. The value for each of the 5 days was averaged.
Time Frame: Days 1 to 5
Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

2. Secondary Outcome: Average Daily Protein Adequacy Over the Study Treatment Period
Description: Average daily protein adequacy received through enteral nutrition is defined as percentage of goal protein delivered per day, where percentage of protein goal delivered is calculated as the ratio of actual protein achievement to the total participant-specific target protein prescribed. The value for each of the 14 days was averaged.
Time Frame: Days 1 to 14
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Average Daily Change in 24-hour Gastric Residual Volume (GRV) Over the First 5 Days of Study Treatment
Description: GRV is defined as the volume of fluid remaining in the stomach at a point in time during enteral nutrition feeding. The value for each of the 5 days was averaged.
Time Frame: Days 1 to 5
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Average Daily Caloric Adequacy
Description: Average daily caloric adequacy received through enteral nutrition was defined by percentage of goal calories achieved per day (percentage calorie goal achieved=actual calorie achievement/total participant-specific target calories). The values in the 5-day period and the 14-day period were averaged.
Time Frame: Days 1 to 5 and Days 1 to 14
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Resolution of Enteral Feeding Intolerance (EFI)
Description: Time to resolution of EFI is defined as the time needed to achieve GRV less than or equal to 250 ml in the absence of vomiting/retching.
Time Frame: Days 1 to 14 or until resolution of EFI, whichever occurs first
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Achieving at Least 80% of Daily Goal Calories
Time Frame: Days 1 to 14 or end of treatment
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants Achieving at Least 80% of Daily Goal Protein
Time Frame: Days 1 to 14 or end of treatment
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Ctrough: Observed Concentration at the End of a Dosing Interval of TAK-954
Time Frame: Day 5 pre-dose
Population: as for outcome 1
Arm/Group | TAK-954 0.1 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Arm/Group | TAK-954 0.1 mg
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03477903/Prot_SAP_000.pdf